CLINICAL TRIAL: NCT02447484
Title: Texting Intervention to Sustain HIV Prevention in Women in High-drug-use Contexts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Comisión de Salud Fronteriza México-Estados Unidos (CSFMEU) (Unknown)
Responsible Party: Principal Investigator, Thomas L. Patterson, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01DA039071 (NIH)
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: HIV; Syphilis; Gonorrhea; Chlamydia
Keywords: female sex workers; HIV sexual risk reduction; behavior maintenance; text messaging
MeSH Terms: conditions — Syphilis; Gonorrhea; Chlamydia Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mujer Segura Siempre (Experimental): Twice-daily safer-sex and safer-drug-use text messages, 5 days per week, for 24 months. Text message content based on 8 different constructs of behavior-maintenance theory and tailored to specific preferences and motivators provided by participant.
  Interventions: Behavioral: Mujer Segura Siempre
- General Health Message Texts (Active Comparator): Twice-daily text messages, 5 days per week, for 24 months. Text message content centered on general health promotion, including getting regular medical checkups and maintaining good dietary and exercise habits.
  Interventions: Behavioral: General Health Message Texts

INTERVENTIONS:
Behavioral: Mujer Segura Siempre — Participants receive personalized text messages twice a day, five days per week. Messages are designed to encourage women to maintain positive behavioral changes they have made in response to the baseline safer-sex training that is delivered to all participants regardless of intervention assignment. Message content is based upon theoretical constructs of behavior-change maintenance as articulated by Voils et al. (Health Education & Behavior, 2013). Personalization elements include participant's name, times of day when she prefers to receive messages, and specific motivators of behavior change she expressed in the baseline interview.
  Arms: Mujer Segura Siempre
Behavioral: General Health Message Texts — Participants receive generic health-promotion text messages twice a day, five days per week.
  Arms: General Health Message Texts

SUMMARY:
The purpose of this study is to determine whether a program of regular, theory-based text messages that encourages the message recipient to continue practicing safer sex (i.e., using condoms with sex partners) is effective in maintaining positive behavior change in women who have completed a brief safer-sex training.

DETAILED DESCRIPTION:
The overarching aim of this study is to evaluate the efficacy of a technology-enabled behavioral intervention, Mujer Segura Siempre (Healthy Woman Forever: MSS), that is designed to maintain the effects of a brief, single-session sexual risk reduction intervention (Mujer Más Segura: MMS) that was proven efficacious in reducing incidence of HIV and sexually transmitted infections (STIs) among drug- and non-drug-using Mexican female sex workers (FSWs) in Tijuana and Ciudad Juarez. Despite the efficacy of MMS, it is well known that treatment effects of health behaviors erode and that adherence to new health behaviors is often poor, with relapse rates up to 50% or more within 6 months, perhaps because the constructs responsible for behavior acquisition differ from those that sustain behavior change. This innovative behavior-maintenance intervention, Mujer Segura Siempre (MSS), will be delivered using text messaging. It incorporates concepts that are theorized to be important to sustain positive behavior change, and it builds on maintenance-specific content and skills that have been significant in interventions focused on other health behaviors (e.g., smoking cessation, weight loss). All women enrolled in the study will begin by receiving the Mujer Más Segura (MMS) counseling, with specific information for women who are intravenous drug users (IDU) in addition to being FSWs. High levels of injection and non-injection drug use have been reported by FSWs and their male clients in our study sites, making it imperative to address safer injection practices in both the initial behavior change program and in our text-based maintenance program.

The text messages that constitute the experimental part of this study will be based on maintenance-specific behavioral and cognitive constructs that are theorized to be involved in behavior maintenance, including self-regulatory focus, maintenance self-efficacy, and relapse prevention planning. The MSS text messaging maintenance intervention will be compared to time-equivalent exposure to general health text messages. Our specific aims are:

Aim 1: Determine if the MSS intervention (MMS counseling plus 24 months of behavioral maintenance text messages-Group 1) is associated with significant reductions in HIV/STI incidence (primary outcome) relative to a time-equivalent control condition (counseling + 24 months of general health text messages-Group 2) among drug-using and non-drug-using FSWs in Tijuana and Cd. Juarez.

Aim 2: Determine if the MSS intervention is associated with increased use of condoms for vaginal and anal sex with male clients, better attendance at regularly scheduled STI screenings, and reduced sharing of injection equipment for FSW-IDU (secondary outcomes) relative to a time-equivalent control condition.

Aim 3: Determine if substance use factors (frequency, intensity, and patterns of alcohol and drug use, including injection use, binge use, polydrug use) mediate or moderate intervention efficacy, taking into account structural and environmental risk factors (e.g., availability of condoms, drugs in the workplace), maintenance constructs (e.g., relapse prevention planning, self-efficacy maintenance), and personal characteristics (e.g., age, sexual abuse, depression).

Aim 4: Evaluate the cost-effectiveness of MSS compared to the control condition, Mujer Más Segura alone (based on data from previous studies), and usual care in Mexico.

To accomplish these aims, investigators will deliver MSS to 600 HIV-negative FSWs (300 in Tijuana, 300 in Cd. Juarez) who report unsafe sex with at least one client in the previous 6 months, and randomize them to either one of two groups: Group 1 (n=300), MSS text-based maintenance program for 24 months post-counseling; or Group 2 (control condition, n=300) general health text messages for 24 months post counseling. Both groups will be assessed at 6, 12, 18, and 24 months post-counseling.

ELIGIBILITY:
Inclusion Criteria:

* Biologically female,
* at least 18 years old,
* report having exchanged sex for money, goods, shelter or drugs within the previous 30 days,
* test HIV-negative at baseline,
* agreeable to receiving antibiotic treatment for chlamydia, gonorrhea, syphilis and trichomoniasis if they test positive (to allow us to differentiate incident from prevalent cases at follow-up),
* report having unprotected vaginal or anal sex with a male client at least once during the previous month, and
* be treatment-naive (i.e., must not have already participated in the Mujer Segura or Mujer Más Segura safer-sex interventions).

Exclusion Criteria:

* Consistent use of condoms for vaginal and anal sex with all male clients during the previous month,
* known to be HIV+ or test HIV+ for the first time on-site,
* under 18 years of age,
* male or transgendered, and
* incapable of giving informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2015-07-01; Primary Completion 2021-04-30 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
HIV and STI incidence | 24 months

SECONDARY OUTCOMES:
Condom use | 24 months
  Number of times a condom is used expressed as a proportion of total number of vaginal and anal sex acts with male clients
Attendance at regularly scheduled STI screenings | 24 months
  Percentage of regularly scheduled STI screenings that participant attends during the 24-month follow-up period
Sharing of injection equipment | 24 months
  Applies to IDU participants only: number of times participant shared her injection equipment (needles, etc.) with another IDU expressed as a proportion of total number of injection events within a specified recall period

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Patterson, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- PreveCasita, Tijuana, Estado de Baja California, Mexico

REFERENCES:
- [Derived] Patterson TL, Pitpitan EV, Pines HA, Semple SJ, Harvey-Vera A, Depp C, Moore DJ, Martinez G, Rangel MG, Strathdee SA. A Randomized Controlled Trial of a Texting Intervention to Maintain Sexual Risk Reduction with Clients Among Female Sex Workers in Tijuana and Ciudad Juarez, Mexico. AIDS Behav. 2020 Dec;24(12):3306-3319. doi: 10.1007/s10461-020-02930-1. PMID 32444901
- [Derived] Pines HA, Semple SJ, Strathdee SA, Hendrix CW, Harvey-Vera A, Gorbach PM, Magis-Rodriguez C, Martinez G, Patterson TL. Vaginal washing and lubrication among female sex workers in the Mexico-US border region: implications for the development of vaginal PrEP for HIV prevention. BMC Public Health. 2018 Aug 14;18(1):1009. doi: 10.1186/s12889-018-5946-z. PMID 30107833